CLINICAL TRIAL: NCT00006362
Title: A Phase I and Pharmacologic Study of the Proteasome Inhibitor PS-341 in Patients With Advanced Solid Tumors and B-cell Lymphoproliferative Disorders
Brief Title: PS-341 in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Alex A. Adjei, M.D., Mayo Clinic Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000068233; U01CA069912 (NIH); P30CA015083 (NIH); 980111 (Other: Mayo Clinic Cancer Cancer); 1443-99 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Precancerous Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: monoclonal gammopathy of undetermined significance; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; stage III multiple myeloma; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; unspecified adult solid tumor, protocol specific; B-cell chronic lymphocytic leukemia; untreated hairy cell leukemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; primary systemic amyloidosis; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Precancerous Conditions; Monoclonal Gammopathy of Undetermined Significance; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Immunoglobulin Light-chain Amyloidosis; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of PS-341 in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and toxicity of PS-341 in patients with advanced malignancies.
* Determine, in a preliminary manner, the therapeutic activity of this regimen in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

* Regimen A: Patients receive PS-341 IV twice weekly for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of PS-341 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 1 of 3-4 or 2 of 6 patients experience dose-limiting toxicity.

* Regimen B: Once the MTD has been determined in regimen A, patients receive PS-341 IV twice weekly for 2 weeks. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed for 3 months.

PROJECTED ACCRUAL: A maximum of 78 patients will be accrued for this study within 14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven advanced malignancy, including non-Hodgkin's lymphoma (NHL), for which there is no known standard therapy that is potentially curative or definitely capable of extending life expectancy

  * Patients with B-cell lymphoproliferative disorders and a leukemic phase are eligible once the maximum tolerated dose is established
* NHL patients must meet the following conditions:

  * No greater than 25% of bone marrow involved
  * No symptomatic brain metastases
  * Prior brain metastases allowed if definitively treated (radiotherapy and/or surgery) and stable for at least 8 weeks

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST or ALT no greater than 2.5 times ULN (5 times ULN if liver involvement)

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* No uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy or immunotherapy
* No concurrent immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to greater than 30% of bone marrow
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No concurrent antiretroviral therapy (HAART) for HIV positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex A. Adjei, MD, PhD, Study Chair — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin